CLINICAL TRIAL: NCT03072979
Title: Reduction in Tumour Perfusion for Spine Metastasis Treated With Stereotactic Body Radiotherapy (SBRT)
Brief Title: A Study to Quantify Tumour Perfusion for Spine Metastasis Treated With Stereotactic Body Radiotherapy (SBRT)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National University of Singapore (Other)
Responsible Party: Principal Investigator, Radiation Oncology, Dr Balamurugan Vellayappan, National University Hospital, Singapore
Other Study IDs: 2016/01179
Record Dates: First submitted 2017-02-28; First posted 2017-03-08 (Actual); Last update posted 2017-03-08 (Actual); Status verified 2017-03

CONDITIONS: Spine Metastasis
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Stereotactic body radiotherapy — Stereotactic body radiotherapy

SUMMARY:
Pre-clinical evidence suggests that radiotherapy reduces tumour-associated vasculature. The investigators will conduct a single-arm prospective study to quantify the reduction in tumour vasculature post-radiotherapy

ELIGIBILITY:
Inclusion Criteria:

* Age ≥21 years of age
* Proven metastatic disease, excluding haematological and germ cell neoplasms
* Life expectancy >3 months, Eastern Cooperative Oncology group (ECOG) 0-2

Exclusion Criteria:

* The patient must not have an allergy to gadolinium contrast that will limit the ability to image the tumour by MRI safely even with the use of premedication
* eGFR < 30 mL/min or if patient is suffering from acute renal insufficiency
* Prior radiotherapy to the specified region
* Recent surgery to affected spinal levels, or patients requiring immediate surgical intervention
* Spinal instability score (SINS) >12
* Symptomatic cord compression (Bilksy grade 2 or 3), or worsening neurological deficits
* Body weight of more than 120kg
* Pregnancy

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 18 patients from National University Hospital (NUH) will be enrolled. Informed consent will be taken from patients prior to trial entry at NUH.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Estimated)
Dates: Start 2017-01-21 (Actual); Primary Completion 2017-12-31 (Estimated); Study Completion 2018-12-31

PRIMARY OUTCOMES:
Reduction in vasculature | 3 month
  Reduction in vasculature measured by changes on Dynamic Contrast enhanced MRI

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided